CLINICAL TRIAL: NCT01689909
Title: Reducing Suicidal Ideation Through Insomnia Treatment
Acronym: REST-IT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Wake Forest University Health Sciences (Other); University of Wisconsin, Madison (Other); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01MH095776-01A1 (NIH); 1R01MH095776 (NIH)
Record Dates: First submitted 2012-09-18; First posted 2012-09-21 (Estimated); Results first posted 2018-06-20 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Insomnia; Depression; Suicidal Ideation
Keywords: Insomnia; Depression; Suicidal ideation; Zolpidem CR; Placebo
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Suicidal Ideation | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zolpidem-CR (Active Comparator): Zolpidem 6.25 or 12.5 mg in tablet form at nighttime 15 minutes before bed for 8 weeks
  Interventions: Drug: Zolpidem-CR
- Placebo (Placebo Comparator): Placebo in tablet form at nighttime 15 minutes before bed for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zolpidem-CR — Zolpidem 6.25 mg or 12.5 mg in tablet form at nighttime 15 minutes before bed for 8 weeks
  Other Names: Ambien CR
  Arms: Zolpidem-CR
Drug: Placebo — Placebo in tablet form at nighttime 15 minutes before bed for 8 weeks
  Arms: Placebo

SUMMARY:
Epidemiologic reports have linked insomnia to suicidal ideation and suicide death. However, no studies have determined whether treating insomnia decreases the risk of suicidality. We have new data indicating that (1) the link between insomnia and suicidal ideation holds true in clinical trials of depressed insomniacs, (2) dysfunctional cognitions about sleep are related to suicidal ideas, and (3) treatment of insomnia with hypnotics leads to a reduction of suicidal ideation. We now propose to test whether cautious use of hypnotics in suicidal, depressed insomniacs may reduce suicide risk in a multi-site clinical trial.

DETAILED DESCRIPTION:
Primary Aim: We will assess the effect of treating insomnia with hypnotic medication on the intensity of suicidal ideation in depressed outpatients with insomnia and suicidal ideation.

-Hypothesis 1. Treatment of depressed, insomniac and suicidal outpatients with open-label fluoxetine (FLX) and blinded zolpidem controlled release (ZOL) will reduce suicidal ideation more than treatment with FLX and blinded placebo.

Secondary Aim: We will examine whether reduced suicidal ideation in depressed insomniacs is mediated through reduced dysfunctional beliefs about sleep, reduced hopelessness, or fewer nightmares.

* Hypothesis 2a. Reduction in suicidal ideation will be mediated through reductions in dysfunctional beliefs about sleep.
* Hypothesis 2b. Reduction in suicidal ideation will be mediated through reductions in hopelessness.
* Hypothesis 2c. Reduction in suicidal ideation is mediated through fewer nightmares.

Tertiary Aim: We will confirm findings from our prior pilot studies that treatment of insomnia in depressed insomniacs leads to improvements in health-related quality of life, especially in women.

Exploratory Aim: We will archive actigraphy data to permit future examination to confirm our preliminary data that actigraphic activity decreases as suicidal ideation resolves.

Overview of the Need for and Management of a Collaborative Application: The sample sizes required to satisfy the Aims are relatively large, necessitating the pooled recruiting resources of 3 sites. Georgia Regents University (GRU) will serve both as the coordinating/data management site, as well as a recruiting site, with Duke and Wisconsin as recruiting sites. Project management will be coordinated through an Executive Committee of site principal investigators, under the supervision of a Data and Safety Monitoring Board.

Impact on the Field: This application has the potential to change providers' practice in the approach to treating insomnia in depressed patients with mild-moderate suicidal ideation. It may also reveal the mechanisms whereby insomnia increases the risk for suicidal ideation and behavior, and begin to examine whether there is an actigraphic "signature" for reductions in suicidal ideation. When these lessons are applied to the clinical world, they can be applied with low cost.

ELIGIBILITY:
Inclusion Criteria:

* Persons 18-65 years of age
* Persons with confirmed DSM-IV diagnosis of MDE by SCID
* Persons with Research Diagnostic Criteria diagnosis of insomnia
* Persons free of all psychotropic medications for one week before baseline assessment, except that prior FLX treatment will require 4 weeks of abstinence, and MAOIs will require 2 weeks of abstinence.
* Persons with Scale for Suicide Ideation (SSI) scores >2
* Persons with Hamilton Rating Scale for Depression (HRSD24) score >20
* Persons with Mini Mental State Exam (MMSE) score >24
* Persons with Insomnia Severity Index (ISI) score > 7
* Persons with habitual sleep latency > or = 30 minutes or wake time in the middle of the night of > or = 30 minutes, and sleep efficiency < 85%

Exclusion Criteria:

* Non-English speaking, reading, writing persons
* Persons who pose imminent danger to self or others
* Persons with severe suicidal ideation (C-SSRS Suicidal Ideation Score >3)
* Persons with clinical diagnosis of dementia
* Persons with active or past diagnosis of alcohol or substance abuse, bipolar disorder, schizophrenia per the SCID
* Persons who screen positive for moderate-severe sleep apnea (AHI >10) or a prior sleep laboratory-confirmed diagnosis of a primary sleep disorder, such as sleep apnea or periodic limb movement disorder.
* Persons with BMI > 50
* Persons with a self-reported history of napping > 2 times per week (as these are associated with sleep apnea and periodic limb movement disorder in depressed insomniacs)
* Persons who might be harmed by exposure to hypnotics, including pregnant women and patients with respiratory conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2012-12-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William V McCall, MD, MS, Principal Investigator — Augusta University
Locations (4):
- United States (4):
  - Georgia Regents University, Augusta, Georgia
  - Duke University School of Medicine, Durham, North Carolina
  - Wake Forest University School of Medicine, Wake Forest, North Carolina
  - University of Wisconsin- Madison, Madison, Wisconsin

REFERENCES:
- [Derived] McCall WV, Mercado K, Dzurny TN, McCloud LL, Krystal AD, Benca RM, Rosenquist PB, Looney SW. Insomnia and the effect of zolpidem-extended-release on the sleep items of the Hamilton Rating Scale for Depression in outpatients with depression, insomnia, and suicidal ideation: Relationship to patient age. J Psychopharmacol. 2024 Sep;38(9):827-831. doi: 10.1177/02698811241268900. Epub 2024 Aug 9. PMID 39119911
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] McCall WV, Benca RM, Rumble ME, Krystal AD. Blinding and bias in a hypnotic clinical trial. Hum Psychopharmacol. 2021 Jan;36(1):1-5. doi: 10.1002/hup.2757. Epub 2020 Sep 11. PMID 32918323
- [Derived] Rumble ME, McCall WV, Dickson DA, Krystal AD, Rosenquist PB, Benca RM. An exploratory analysis of the association of circadian rhythm dysregulation and insomnia with suicidal ideation over the course of treatment in individuals with depression, insomnia, and suicidal ideation. J Clin Sleep Med. 2020 Aug 15;16(8):1311-1319. doi: 10.5664/jcsm.8508. PMID 32329435
- [Derived] McCall WV, Benca RM, Rosenquist PB, Youssef NA, McCloud L, Newman JC, Case D, Rumble ME, Szabo ST, Phillips M, Krystal AD. Reducing Suicidal Ideation Through Insomnia Treatment (REST-IT): A Randomized Clinical Trial. Am J Psychiatry. 2019 Nov 1;176(11):957-965. doi: 10.1176/appi.ajp.2019.19030267. Epub 2019 Sep 20. PMID 31537089
- [Derived] McCall WV, Benca RM, Rumble ME, Case D, Rosenquist PB, Krystal AD. Prevalence of obstructive sleep apnea in suicidal patients with major depressive disorder. J Psychiatr Res. 2019 Sep;116:147-150. doi: 10.1016/j.jpsychires.2019.06.015. Epub 2019 Jun 19. PMID 31238203

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zolpidem-CR | Placebo
Started | 51 | 52
Completed | 51 | 52
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zolpidem-CR | Placebo | Total
Number analyzed (Participants) | 51 | 52 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 52 | 103
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (14.5) | 41.2 (12.0) | 40.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 19 | 20 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 47 | 51 | 98
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 16 | 28
  White | 34 | 34 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 51 | 52 | 103
Scale for Suicide Ideation [Mean (Standard Deviation); unit: units on a scale] — This is the total score for the Scale for Suicide Ideation. It has 19 items, each scored 0-2, for a maximum of 38 points. Higher scores indicate worse suicidal ideation
  units on a scale | 12.2 (5.3) | 11.8 (5.3) | 12.0 (5.3)
Columbia Suicide Severity Rating Scale (C-SSRS) - suicide ideation scale [Mean (Standard Deviation); unit: units on a scale] — The suicide ideation scale of the C-SSRS is rated 0-5, with "0" meaning no suicidal ideation, "1" meaning a wish to be dead, "2" meaning non-specific active suicidal thoughts, "3" meaning active suicidal ideation with any methods but no plan or intent, "4" meaning active suicidal ideation with some intent but no specific plan, and "5" meaning active suicidal ideation with intent and a specific plan.
  units on a scale | 1.71 (10.3) | 1.58 (10.2) | 1.64 (1.02)
Hamilton Rating Scale for Depression -24 [Mean (Standard Deviation); unit: units on a scale] — This version of the Hamilton Rating Scale for Depression uses 24 items, with a possible total score ranging from 0-74, with higher scores indicating worse depression
  units on a scale | 28.7 (4.7) | 29.6 (7.0) | 29.1 (5.9)
Disturbing Dreams Nightmare Severity Index [Mean (Standard Deviation); unit: units on a scale] — This self-rated scale has 5 items, with asymmetric weighting of each item. The range of the total score is 0-37, with higher scores indicating worse nightmares
  units on a scale | 10.5 (8.8) | 10.2 (7.7) | 10.3 (8.2)
Insomnia Severity Index [Mean (Standard Deviation); unit: units on a scale] — The Insomnia Severity Index is self rated. It has 7 items, each scored 0-4. Therefore the range of scores is 0-28, with higher scores indicating worse insomnia
  units on a scale | 20.6 (3.9) | 21.1 (4.3) | 20.8 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Scale for Suicide Ideation Index (SSI)
Description: This is the total score for the Scale for Suicide Ideation. It has 19 items, each scored 0-2, for a maximum of 38 points. Higher scores indicate worse suicidal ideation
Time Frame: Over 8 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Zolpidem-CR | Placebo
Number analyzed (Participants) | 51 | 52
units on a scale | 4.66 (0.58) | 5.25 (0.59)

2. Primary Outcome: Columbia Suicide Severity Rating Scale (C-SSRS): the Suicidal Ideation Scale
Description: The suicide ideation scale of the C-SSRS is rated 0-5, with "0" meaning no suicidal ideation, "1" meaning a wish t be dead, "2" meaning non-specific active suicidal thoughts, "3" meaning active suicidal ideation with any methods but no plan or intent, "4" meaning active suicidal ideation with some intent but no specific plan, and "5" meaning active suicidal ideation with intent and a specific plan
Time Frame: 8 weeks of treatment
Population: all evaluable randomized participants
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Zolpidem-CR | Placebo
Number analyzed (Participants) | 51 | 52
units on a scale | 0.5447 (0.0869) | 0.8067 (0.0875)

3. Secondary Outcome: Dysfunctional Beliefs and Attitudes About Sleep
Description: The Dysfunctional Beliefs and Attitudes About Sleep scale has 16 items and is self administered. Each item is scored 0-10. The total score is an average of the scores of the 16 items. Hence the range of the total score is also 0-10, with higher scores indicating greater dysfunctional beliefs about sleep
Time Frame: 8 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Zolpidem-CR | Placebo
Number analyzed (Participants) | 51 | 52
units on a scale | 6.03 (0.171) | 6.07 (0.171)

4. Secondary Outcome: Disturbing Dreams and Nightmares Severity Index (DDNSI)
Description: This self-rated scale has 5 items, with asymmetric weighting of each item. The range of the total score is 0-37, with higher scores indicating worse nightmares
Time Frame: 8 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Zolpidem-CR | Placebo
Number analyzed (Participants) | 51 | 52
units on a scale | 5.74 (0.710) | 6.44 (0.718)

5. Secondary Outcome: Beck Hopelessness Scale (BHS)
Description: The Beck Hopelessness Scale is self administered and has 20 'true/false' choices. Some items are reversed scored. The range of scores for the total is 0-20, with higher scores indicating greater hopelessness
Time Frame: 8 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Zolpidem-CR | Placebo
Number analyzed (Participants) | 51 | 52
units on a scale | 9.40 (0.58) | 9.63 (0.58)

6. Secondary Outcome: Hamilton Rating Scale for Depression (HAM-D)
Description: This version of the Hamilton Rating Scale for Depression uses 24 items, with a possible total score ranging from 0-74, with higher scores indicating worse depression
Time Frame: 8 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Zolpidem-CR | Placebo
Number analyzed (Participants) | 51 | 52
units on a scale | 14.93 (0.87) | 15.89 (0.88)

7. Secondary Outcome: Insomnia Severity Index (ISI)
Description: The Insomnia Severity Index is self rated. It has 7 items, each scored 0-4. Therefore the range of scores is 0-28, with higher scores indicating worse insomnia
Time Frame: 8 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Zolpidem-CR | Placebo
Number analyzed (Participants) | 51 | 52
units on a scale | 11.28 (0.62) | 13.72 (0.63)

8. Other Pre Specified Outcome: Basis-32 - the Daily Living and Role Functioning (DLRF) Subscale
Description: This is one of the subscales of the Basis 32. It is self-administered. This subscale has 7 items, each scored 0-4. The totals score is an average of the scores of these 7 items. Higher scores indicate more difficulty with daily living and role functioning.
Time Frame: 8 weeks of treatment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Zolpidem-CR | Placebo
Number analyzed (Participants) | 51 | 52
units on a scale | 1.51 (0.102) | 1.60 (0.102)

9. Other Pre Specified Outcome: Actigraphy
Description: This device measures arm motion over time, reported as "average actigraphic activity Level". The scale is reported as a continuous measure ranging from 0-200, and reported as the average score for each hour for all 24-hours of the day. Higher score represent greater c=activity at that point in time
Time Frame: 8 weeks of treatment
Population: participants with depression, insomnia, and suicidality
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Scale for Suicide Ideation Score Greater Than or Equal to 6: Participants with a baseline Scale for Suicide Ideation Score Greater than or Equal to 6
- Scale for Suicide Ideation Score Less Than 6: Participants with Scale for Suicide Ideation Score less than 6
Arm/Group | Scale for Suicide Ideation Score Greater Than or Equal to 6 | Scale for Suicide Ideation Score Less Than 6
Number analyzed (Participants) | 37 | 23
units on a scale | 150 (30) | 170 (30)

ADVERSE EVENTS:
Time Frame: 8 weeks randomized care and 2 weeks of follow up after the end of randomized care
Arm/Group | Zolpidem-CR | Placebo
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/52
Serious Adverse Events (participants affected / at risk) | 1/51 | 0/52
Other Adverse Events (participants affected / at risk) | 31/51 | 37/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zolpidem-CR (N=51) | Placebo (N=52)
pregnancy then miscarriage (Pregnancy, puerperium and perinatal conditions) | 1 | 0 — Despite being cautioned about the need for birth-control, a female participant nevertheless became pregnant (by her report), and shortly thereafter miscarried (by her report). She had a history of multiple prior miscarriages.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zolpidem-CR (N=51) | Placebo (N=52)
cold symptoms and flu (Respiratory, thoracic and mediastinal disorders) | 12 (21) | 9 (9)
nausea and diarrhea (Gastrointestinal disorders) | 9 (14) | 9 (14)
headache (Nervous system disorders) | 6 (9) | 6 (11)
Other (General disorders) | 4 (14) | 13 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT01689909/Prot_SAP_000.pdf